CLINICAL TRIAL: NCT02789865
Title: Multicenter Prospective Randomized Clinical Trial Comparing Endoscopic Retrograde Appendicitis Therapy (ERAT) vs Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis
Brief Title: Clinical Trial Comparing ERAT vs Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 3201 Hospital in Hanzhong (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-010
Record Dates: First submitted 2016-04-24; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Acute Appendicitis
Keywords: Acute appendicitis; Endoscopic retrograde appendicitis therapy; Endoscopic retrograde appendicography; Endoscopic therapy; Appendectomy; Antibiotic Therapy
MeSH Terms: conditions — Appendicitis | interventions — Ertapenem; Levofloxacin; Metronidazole; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Antibiotic therapy group (Active Comparator): The patients will be treated with intravenous broad-spectrum antibiotics (Ertapenem 1g/d) for 3 days and oral antibiotics (Levofloxacin 500mg once daily and Metronidazole 500mg 3 times per day) for 7 days. If patients in the antibiotic group deteriorate during the hospital stay (suspicious perforation or any symptoms of peritonitis) patients will be operated.
  Interventions: Drug: Ertapenem, Levofloxacin and Metronidazole
- ERAT group (Experimental): The patients will receive emergent endoscopic retrograde appendicitis therapy (ERAT).
  Interventions: Procedure: Endoscopic retrograde appendicitis therapy (ERAT)
- Appendectomy group (Active Comparator): The patients will receive laparoscopic appendectomy according to standard routines.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Drug: Ertapenem, Levofloxacin and Metronidazole — The patients will be treated with intravenous broad-spectrum antibiotics (Ertapenem 1g/d) for 3 days and oral antibiotics (Levofloxacin 500mg once daily and Metronidazole 500mg 3 times per day) for 7 days. If patients in the antibiotic group deteriorate during the hospital stay (suspicious perforation or any symptoms of peritonitis) patients will be operated.
  Arms: Antibiotic therapy group
Procedure: Endoscopic retrograde appendicitis therapy (ERAT) — The procedures of ERAT will be performed as below：1.Cannulation of the appendiceal lumen. 2.Endoscopic retrograde appendicography (ERA). 3.Irrigation and appendicolith removal. 4.Stenting for drainage.
  Arms: ERAT group
Procedure: Appendectomy — The patients will receive laparoscopic appendectomy according to standard routines.
  Arms: Appendectomy group

SUMMARY:
Endoscopic retrograde appendicitis therapy (ERAT) is a new and minimally invasive method for the diagnosis and treatment of acute appendicitis.After a positive diagnosis of acute appendicitis is established by either colonoscopic direct-vision imaging or fluoroscopic endoscopic retrograde appendicography (ERA) imaging in patients with suspected acute appendicitis, the procedures to relieve the appendiceal lumen obstruction including appendiceal luminal irrigation, appendicolith removal, and stenting for drainage whenever necessary will be carried out. In this multicenter prospective randomized clinical trial, the patients with uncomplicated acute appendicitis will be divided into three groups randomly: ERAT group, antibiotic therapy group and appendectomy group. The primary outcome is duration of abdominal pain. The secondary outcomes include mean hospital stay, mean operative time, duration of fever, duration of leukocytosis, bed time, rate of complication, rate of recurrence and rate of appendectomy during follow-up period of 1 year.

DETAILED DESCRIPTION:
Intervention

The patients with uncomplicated acute appendicitis will be divided into three groups randomly: ERAT group, antibiotic therapy group and appendectomy group.

1) ERAT group: In preparation for ERAT, low-pressure cleansing enemas (500 mL normal saline solution per enema) will be administered for three times before the procedures for bowel preparation. Antibiotic therapy (levofloxacin + metronidazole) will be intravenously administrated to the patients in the perioperative period.

The procedures of ERAT will be performed as below：

1. Cannulation of the appendiceal lumen: Colonoscopic examination under direct vision of the whole colon, ileocecal junction and terminal ileum will be performed to exclude other abnormalities first, and focus on the appendiceal orifice and the surrounding mucosa. Colonoscope attached by a transparent cap will be positioned close to the appendiceal oriﬁce. Gerlach's valve will be pushed aside using the transparent cap, a standard catheter loaded with a 0.035-inch guidewire (loop-tip or hydrophilic-tip) will be placed in the appendiceal oriﬁce. The guidewire will be probed gently to insert into the appendiceal lumen. The catheter will be then subsequently moved forward after the guidewire inserting deeply into the lumen under fluoroscopic guidance.
2. Endoscopic retrograde appendicography (ERA): After cannulation of the appendiceal lumen, decompression of lumen will be achieved by suction using a 5-mL syringe attached to the catheter. A soluble contrast agent (iobitridol) will be then used to fill the appendix while being monitored by fluoroscopy to check the radiographic features of the appendix (including position, length, contour, mobility, intraluminal content and inner diameter of appendiceal lumen).
3. Irrigation and appendicolith removal: The appendiceal lumen will be irrigated with normal saline solution to clear away the pus and the sand-like appendicoliths, while the large appendicoliths will be extracted using a balloon catheter or an extraction basket.
4. Stenting for drainage: If the pus is massive or the lumen is stenosis, a plastic straight stent (8.5F) will be placed into the lumen over the guidewire for luminal decompression with the plan to retrieve the stent after about one week.

2) Antibiotic therapy group: The patients will be treated with intravenous broad-spectrum antibiotics (Carbapenems) for 3 days and oral antibiotics (Levofloxacin and Metronidazole) for 7 days. If patients in the antibiotic group deteriorate during the hospital stay (suspicious perforation or any symptoms of peritonitis) patients will be operated.

3) Appendectomy group: The patients will undergo laparoscopic appendectomy according to standard routines.

Follow-up and outcome measures

Follow-up will be performed until the end of the study period. The primary outcome is duration of abdominal pain. The secondary outcomes include mean hospital stay, mean operative time, duration of fever, duration of leukocytosis, bed time, rate of complication, rate of recurrence and rate of appendectomy during follow-up period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with Alvarado scores ≥7 (with or without US/CT) diagnosed of uncomplicated acute appendicitis
* patients with Alvarado scores <7 but US/CT suggested uncomplicated acute appendicitis or could not exclude acute appendicitis.

Exclusion Criteria:

* perforated appendicitis
* periappendiceal abscess
* contraindications for colonoscopy
* allergy to contrast media or iodine
* pregnancy
* unable to cooperate or provide informed consent

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
duration of abdominal pain | up to 10 days

SECONDARY OUTCOMES:
mean hospital stay | up to 10 days
duration of fever | up to 10 days
duration of leukocytosis | up to 10 days
bed time | up to 10 days
rate of complication | during follow-up period of 1 year
rate of recurrence | during follow-up period of 1 year
rate of appendectomy | during follow-up period of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yingchao Li, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (3):
- China (3):
  - 3201 Hospital of Hanzhong, Hanzhong, Shaanxi
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vons C, Barry C, Maitre S, Pautrat K, Leconte M, Costaglioli B, Karoui M, Alves A, Dousset B, Valleur P, Falissard B, Franco D. Amoxicillin plus clavulanic acid versus appendicectomy for treatment of acute uncomplicated appendicitis: an open-label, non-inferiority, randomised controlled trial. Lancet. 2011 May 7;377(9777):1573-9. doi: 10.1016/S0140-6736(11)60410-8. PMID 21550483
- [Background] Salminen P, Paajanen H, Rautio T, Nordstrom P, Aarnio M, Rantanen T, Tuominen R, Hurme S, Virtanen J, Mecklin JP, Sand J, Jartti A, Rinta-Kiikka I, Gronroos JM. Antibiotic Therapy vs Appendectomy for Treatment of Uncomplicated Acute Appendicitis: The APPAC Randomized Clinical Trial. JAMA. 2015 Jun 16;313(23):2340-8. doi: 10.1001/jama.2015.6154. PMID 26080338
- [Background] Liu BR, Ma X, Feng J, Yang Z, Qu B, Feng ZT, Ma SR, Yin JB, Sun R, Guo LL, Liu WG. Endoscopic retrograde appendicitis therapy (ERAT) : a multicenter retrospective study in China. Surg Endosc. 2015 Apr;29(4):905-9. doi: 10.1007/s00464-014-3750-0. Epub 2014 Aug 9. PMID 25106722